CLINICAL TRIAL: NCT04776642
Title: "Arrhythmia and Conduction Disorders: TowArd Pathophysiology Based Treatment" ADAPT Biobank
Brief Title: Biobank for "Arrhythmia and Conduction Disorders: TowArd Pathophysiology Based Treatment"
Acronym: ADAPT
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.R. de Groot, Prof.dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2014_054#A201436
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Arrythmia; Conduction Disorder; Pathophysiology
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Biological Specimen Banks; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * left atrial appendage tissue
  * blood
  * one or more of following fat patches: epicardial fat, subcutaneous fat, pericardial fat, visceral fat.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- MARK_AF: MARKers of ATrial Remodeling in Patietns with Atrial Fibrillation. Patients with paroxysmal and persistent atrial fibrillation undergoing thoracoscopic atrial fibrillation ablation surgery
  Interventions: Other: Biobank for Left atrial appendage tissue; Other: Biobank for Blood; Other: Biobank for One or more of following fat patches: epicardial fat, subcutaneous fat, pericardial fat, visceral fat.
- INDICO AF: Atrial Fibrillation in Patients With an Implantable Cardioverter Defibrillator and Coronary Artery Disease. Investigate the incidence of new-onset AF in patients with coronairy artery disease and an impaired LVEF, who will receive a single chamber ICD as primary prevention for sudden cardiac death.
  Interventions: Other: Biobank for Blood
- PREDICT AF: PREDICT AF, Tissue, Blood and biomarkers to predict future Atrial Fibrillation. Patients without a history of atrial fibrillation undergoing cardiothoracic surgery
  Interventions: Other: Biobank for Left atrial appendage tissue; Other: Biobank for Blood; Other: Biobank for One or more of following fat patches: epicardial fat, subcutaneous fat, pericardial fat, visceral fat.
- WEIGHTLOSS AF: The change of adipose tissue characteristics upon drastic weight loss: Implications for atrial fibrillation.
  Interventions: Other: Biobank for Blood; Other: Biobank for One or more of following fat patches: epicardial fat, subcutaneous fat, pericardial fat, visceral fat.
- MAD AF: (123I-mIBG And Defibrillation for Atrial Fibrillation) Enhanced sympathetic activity as a mechanism of Atrial Fibrillation. Patients will undergo 123I-mIBG scintigraphy within 7 days before and six week after an elective cardioversion is performed.
  Interventions: Other: Biobank for Blood
- Adapt Biobank - AF surgery: Patients with Atrial Fibrillation who only donate blood and tissue for the biobank. Patients undergo thorascopic surgery, LAA will be amputated, blood will be collected.
  Interventions: Other: Biobank for Left atrial appendage tissue; Other: Biobank for Blood; Other: Biobank for One or more of following fat patches: epicardial fat, subcutaneous fat, pericardial fat, visceral fat.
- Adapt Biobank - blood: Patients with cardiac arrhythmias who only donate blood for the ADAPT biobank.
  Interventions: Other: Biobank for Blood

INTERVENTIONS:
Other: Biobank for Left atrial appendage tissue — Bodily material is used for biochemical marker assessments, histological and molecular analyses for research in cardiac arrhythmias.
  Groups: Adapt Biobank - AF surgery; MARK_AF; PREDICT AF
Other: Biobank for Blood — Bodily material is used for biochemical marker assessments, histological and molecular analyses for research in cardiac arrhythmias.
Other: Biobank for One or more of following fat patches: epicardial fat, subcutaneous fat, pericardial fat, visceral fat. — Bodily material is used for biochemical marker assessments, histological and molecular analyses for research in cardiac arrhythmias.
  Groups: Adapt Biobank - AF surgery; MARK_AF; PREDICT AF; WEIGHTLOSS AF

SUMMARY:
The 'ADAPT' Biobank is a collection of body material and data from patients with or at risk of cardiac arrhythmias who underwent or will undergo (non-) invasive treatment for this disease. Its main objective is to obtain a comprehensive collection of patient information and material to facilitate research and gain better insight into the complex pathophysiology of the different arrhythmias, the multifactorial process, the heterogeneity in clinical presentation, and prognosis.

Bodily material is used for biochemical marker assessments, histological and molecular analyses for research in cardiac arrhythmias.

DETAILED DESCRIPTION:
The pathophysiological process of many cardiac arrhythmias is complex because of its multifactorial character. Despite extensive research that has already been performed in the field of electrophysiology the exact pathophysiological process of the different arrhythmias remains incompletely understood. The ability to identify subgroups of patients within a population with the same type of arrhythmia that can benefit from a specific treatment strategy might provide more individualized therapeutic opportunities, improve prognostication or provide preventive opportunities in patient with cardiac arrhythmias. Biobanks can make a valuable contribution to the development of diagnostic, preventive and therapeutic methods. More insights into the correlations between genes, environmental factors and susceptibility to illness may be of great value. The 'ADAPT' Biobank has been designed to establish a systematic and qualitative collection of bodily materials for future research in the cardiovascular field. The Biobank includes bodily material of patients with cardiac arrhythmias undergoing (non-) invasive treatment or control patients undergoing cardiothoracic surgery. Clinical data related to the cardiac arrhythmic disease is recorded. The data and samples will be linked to the participants' medical records to allow longitudinal follow-up.

ELIGIBILITY:
Inclusion criteria:

* Patients visiting the AMC outpatient clinic
* Patients included in an ongoing clinical trial linked to this biobank. Studies are listed under point "Groups and interventions" and include:

  * MARK AF
  * INDICO AF
  * PREDICT AF
  * WEIGHTLOSS AF
  * MAD AF
* Patients included in future clinical trial linked to this biobank. Studies may be linked to this biobank that investigates prevalent or incident cardiac arrhythmias.
* Cardiac arrhtymias are defined as

  * Supraventricular tachycardia, among which the most common are:

    * Atrial Fibrillation (AF)
    * Atrial Tachycardia (AT)
    * Atrial Flutter (AFL)
    * Atrioventricular Nodal Reentrant Tachycardia (AVNRT)
    * Atrioventricular Reentrant Tachycardia (AVRT)
  * Ventricular tachycardia, among which the most common are:

    * Ventricular Tachycardia (VT)
    * Ventricular Flutter (VFL)
    * Ventricular Fibrillation (VF)
  * Bradycardia:

    * Sinus Node Dysfunction
    * AV Node Dysfunction
    * Interventricular Conduction Disorder
  * Arrhythmogenic cardiomyopathies, among which the most common are:

    * Dilated Cardiomyopathy
    * Restrictive Cardiomyopathy
    * Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)

Exclusion criteria (shared for all studies):

* Age < 18
* Unable or unwilling to comply with study procedures
* Pregnancy or of childbearing potential without adequate contraception
* NYHA class IV heart failure symptoms or left ventricular ejection fraction <35%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cardiac arrhythmia and are treated in the AMC Heart Center are eligible to donate blood or other bodily material for the 'ADAPT' Biobank. Patient are asked to participate in the 'ADAPT' Biobank during outpatient clinic visits or prior to treatment for their arrhythmia.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-12-18 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
(new onset) atrial fibrilation | 5 year follow up
  obtain a comprehensive collection of patient information and material to facilitate research and gain better insight into the complex pathophysiology of the different arrhythmias
recurrence of cardia arrythmia | 5 year follow up
  obtain a comprehensive collection of patient information and material to facilitate research and gain better insight into the complex pathophysiology of the different arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Joris de Groot, MD, PhD, Principal Investigator — Amsterdam UMC - AMC
Locations (1):
- Amsterdam University Medical Center location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No